CLINICAL TRIAL: NCT03575793
Title: A Phase I/II Study of Nivolumab, Ipilimumab and Plinabulin in Patients With Recurrent Small Cell Lung Cancer: Big Ten Cancer Research Consortium. BTCRC-LUN17-127
Brief Title: A Phase I/II Study of Nivolumab, Ipilimumab and Plinabulin in Patients With Recurrent Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Salma Sabbour (Other)
Collaborators: BeyondSpring Pharmaceuticals Inc. (Industry); Bristol-Myers Squibb (Industry); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor-Investigator, Salma Sabbour, Sponsor Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-LUN17-127
Record Dates: First submitted 2018-06-20; First posted 2018-07-03 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer; SCLC
MeSH Terms: conditions — Lung Neoplasms | interventions — Nivolumab; NPI 2358; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I (Dose Escalation): nivolumab, ipilimumab and plinabulin (Experimental): On Day 1 in a 21-day cycle, all patients will receive nivolumab (1 mg/kg, IV), ipilimumab (3 mg/kg, IV) and plinabulin (escalating cohorts, IV).
  After 4 treatment cycles, ipilimumab will be discontinued and patients will continue treatment with nivolumab 240 mg and plinabulin every 2 weeks (maintenance period) until one of the end of treatment criteria occur.
  Plinabulin escalation is as follows:
  Level -1 : 13.5mg/m^2
  Level 1 (start) : 20mg/m^2
  Level 2 : 30mg/m^2
  Interventions: Drug: Nivolumab; Drug: Plinabulin; Drug: Ipilimumab
- Phase II: nivolumab, ipilimumab, and plinabulin (Experimental): On Day 1 in a 21-day cycle, all patients will receive nivolumab (1 mg/kg, IV), ipilimumab (3 mg/kg, IV) and plinabulin (MTD from Phase I).
  After 4 treatment cycles, ipilimumab will be discontinued and patients will continue treatment with nivolumab 240 mg and plinabulin every 2 weeks (maintenance period) until one of the end of treatment criteria occur .
  Interventions: Drug: Nivolumab; Drug: Plinabulin; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — A fully human immunoglobulin (Ig) G4 monoclonal antibody directed against the negative immunoregulatory human cell surface receptor programmed death-1 (PD-1,PCD-1,) with immune checkpoint inhibitory and antineoplastic activities.
  Other Names: Opdivo
Drug: Plinabulin — Plinabulin (BPI-2358) is a synthetic, low molecular weight, new chemical entity originally developed by Nereus Pharmaceuticals, Inc., and now by BeyondSpring Pharmaceuticals, Inc. It belongs to the diketopiperazine class of compounds with a chemical name 2, 5-piperazinedione, 3-[[5-(1,1-dimethylethyl)-1H-imidazol-4-yl[methylene]-6-(phenylmethylene)-, (3Z,6Z) (trivial name t-butyl-dehydrophenylahistin).
Drug: Ipilimumab — Ipilimumab is a monoclonal antibody that works to activate the immune system by targeting CTLA-4, a protein receptor that downregulates the immune system.
  Other Names: Yervoy

SUMMARY:
This is an open-label Phase I/II study, with a dose escalation part (Phase I) and a single-arm part (Phase II), in patients with recurrent SCLC who progressed after first-line platinum-based chemotherapy and who are candidates for second line therapy. No PK evaluation is planned in this study as nivolumab and ipilimumab are unlikely to alter plinabulin's PK, since the route of excretion is different.

DETAILED DESCRIPTION:
This is an open-label Phase I/II study, with a dose escalation part (Phase I) and a single arm part (Phase II), in patients with recurrent SCLC.

In the Phase I part, patients will receive plinabulin at escalating doses in combination with nivolumab and ipilimumab. Doses of study drug will be administered as intravenous (IV) infusions in 21 day cycles. Patients will receive all study drugs on Day 1 of each cycle. After 4 treatment cycles, ipilimumab is stopped and patients continue treatment with nivolumab and plinabulin every 2 weeks (maintenance period) or until disease progression, development of unacceptable toxicity or one of the protocol-defined reasons for treatment discontinuation occurs.

At least 3 patients will be enrolled in each cohort, starting at 20 mg/m2 of plinabulin. The dose of plinabulin will be escalated in sequential patient cohorts after the safety data from the first cycle is reviewed. Thereafter the dose of plinabulin will be escalated to 30 mg/m2, provided that dose-limiting toxicities (DLTs) are not observed per the specified criteria, until the RP2D is determined.

In the Phase II part, up to 26 patients will be treated with the triple combination of plinabulin (at RP2D) + nivolumab + ipilimumab. Patients will continue treatment until disease progression, development of unacceptable toxicity or one of the protocol-defined reasons for treatment discontinuation occurs.

ELIGIBILITY:
Inclusion Criteria:

The patients must satisfy all of the following inclusion/exclusion criteria in order to be eligible for the study:

* Must have signed and dated written informed consent form in accordance with regulatory and institutional guidelines.
* Males and females aged >18 years at time of consent.
* Histological or cytological confirmed extensive-stage SCLC
* Patients who progressed after at least 1 platinum-based chemotherapy regimen. Patients with platinum resistance (defined as recurrence or progression of disease within 90 days of completion of the platinum-based regimen) are eligible. For phase II, patients also must have been treated with at least one prior line of PD-1/PD-L1 therapy.
* Measurable disease according to RECIST v1.1 (Section 8) obtained by imaging within 28 days prior to study registration.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 14 days before registration and minimum life expectancy of at least 12 weeks.
* Treatment to be initiated at least 2 weeks since last dose of prior systemic anticancer therapy (chemotherapy, radiation, and/or surgery.
* Recovery to grade 1 of any clinically significant toxicity (excluding alopecia, grade 2 fatigue, vitiligo, endocrinopathies on stable replacement therapy) prior to initiation of study drugs.
* Female patients of childbearing potential have a negative pregnancy test at baseline. Females of childbearing potential are defined as sexually mature women without prior hysterectomy or who have had any evidence of menses in the past 12 months. However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti estrogens, or ovarian suppression.

  * Women of childbearing potential (i.e., menstruating women) must have a negative urine pregnancy test (positive urine tests are to be confirmed by serum test) documented within 14 days of study registration and within the 24-hour period prior to the first dose of study drug.
  * Sexually active women of childbearing potential enrolled in the study must agree to use 2 forms of accepted methods of contraception during the course of the study and for 23 weeks after their last dose of study drug. Effective birth control includes (a) intrauterine device plus 1 barrier method; (b) on stable doses of hormonal contraception for at least 3 months (e.g., oral, injectable, implant, transdermal) plus one barrier method; (c) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm); or (d) a vasectomized partner.
  * For male patients who are sexually active and who are partners of premenopausal women: agreement to use 2 forms of contraception as in criterion 9b above during the treatment period and for 31 weeks after the last dose of study drug.
* Adequate laboratory values.

  * Absolute neutrophil count ≥1,000/µL
  * Platelet count ≥100,000/µL
  * Hemoglobin ≥9.0 g/dL
  * Total bilirubin ≤1.5 x upper limit of normal (ULN) or ≤3 x ULN for subjects with Gilbert's disease
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 x ULN (≤5 x ULN if evidence of hepatic involvement by malignant disease)
  * Creatinine ≤ 1.5 x ULN or estimated glomerular filtration rate (eGFR) ≥40 mL/min/1.73m2
  * Lipase and Amylase ≤1.5 x ULN. Subjects with Lipase >1.5 x ULN may enroll if there are neither clinical nor radiographic signs of a pancreatitis.

Exclusion Criteria

Patients with any of the following will be excluded from participation in the study.

* Active interstitial lung disease (ILD) or pneumonitis or a history of ILD or pneumonitis requiring treatment with steroids. Prior history of radiation pneumonitis is allowed if pneumonitis was restricted to the field of radiation.
* History of ileus or other significant gastrointestinal disorder known to increase the risk of ileus or chronic bowel hypomotility
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 23 weeks (female) or 31 weeks (male) after the last dose of study drug.
* Must not have received CTLA-4 targeted therapy previously
* Treatment with any investigational agent within 28 days prior to registration for protocol therapy. Vaccination for SARS-CoV-2 is allowed as well as any therapy as required for the treatment of active COVID 19 infection.
* Known active symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with neurological symptoms must undergo a head computed tomography (CT) scan or brain magnetic resonance imaging (MRI) to exclude brain metastasis. Patients whose brain metastases have been treated may participate provided there is no evidence of progression for at least 2 weeks after CNS-directed treatment, as ascertained by clinical examination or brain imaging.
* Known history of human immunodeficiency virus (HIV) or active hepatitis B (by surface antigen expression or polymerase chain reaction [PCR]) or active hepatitis C (by PCR) infection. NOTE: HIV testing is not required; Hepatitis B and C testing are required at screening.
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to study registration.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs) or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Vitiligo, alopecia, hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment, celiac disease controlled by diet alone or conditions not expected to recur in the absence of an external trigger are permitted.
* A condition requiring systemic treatment with corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to administration of study drugs.
* History of psychiatric illness or social situations that would limit compliance with study requirements. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
* Prior malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) unless a complete remission was achieved at least 2 years prior to study entry.
* Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association (NYHA) Class III-IV within 6 months prior to their first dose of study drugs.
* Evidence of ongoing inadequately controlled hypertension (defined as baseline systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg).
* Any active grade 3 or higher viral, bacterial, or fungal infection within 2 weeks of the first dose of the study drugs. Routine antimicrobial prophylaxis is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salma Jabbour, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Illinois Cancer Center, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Erlanger Health System, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Plinabulin 20mg/m^2 With Nivolumab and Ipilimumab: On Day 1 in a 21-day cycle, all patients will receive nivolumab (1 mg/kg, IV), ipilimumab (3 mg/kg, IV) and plinabulin (20mg/m2, IV) for the first 4 cycles.
  After 4 treatment cycles, ipilimumab will be discontinued and patients will continue treatment with nivolumab 240 mg and plinabulin every 2 weeks (maintenance period) until one of the end of treatment criteria occur.
- Plinabulin 30mg/m^2 With Nivolumab and Ipilimumab: On Day 1 in a 21-day cycle, all patients will receive nivolumab (1 mg/kg, IV), ipilimumab (3 mg/kg, IV) and plinabulin (30mg/m2, IV) for the first 4 cycles.
  After 4 treatment cycles, ipilimumab will be discontinued and patients will continue treatment with nivolumab 240 mg and plinabulin every 2 weeks (maintenance period) until one of the end of treatment criteria occur.
Period: Overall Study
Arm/Group | Plinabulin 20mg/m^2 With Nivolumab and Ipilimumab | Plinabulin 30mg/m^2 With Nivolumab and Ipilimumab
Started | 8 | 31
Completed | 8 | 28
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Never Treated | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plinabulin 20mg/m^2 With Nivolumab and Ipilimumab | Plinabulin 30mg/m^2 With Nivolumab and Ipilimumab | Total
Number analyzed (Participants) | 8 | 28 | 36
Age, Continuous [Median (Full Range); unit: years] | 56.50 [43 to 78] | 64 [43 to 80] | 60 [43 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 17
  Male | 3 | 16 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 7 | 25 | 32
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 8 | 26 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 28 | 36
Brain Metastases [Count of Participants; unit: Participants]
  Yes | 3 | 10 | 13
  No | 5 | 18 | 23
Prior PD-L1 [Count of Participants; unit: Participants] — Programmed Cell Death Ligand 1 (PD-L1) is a trans-membrane protein that is considered to be a co-inhibitory factor of the immune response, it can combine with PD-1 to reduce the proliferation of PD-1 positive cells, inhibit their cytokine secretion and induce apoptosis. PD-L1 also plays an important role in various malignancies where it can attenuate the host immune response to tumor cells.
  Participants
    Prior PD-L1 = Yes | 3 | 27 | 30
    Prior PD-L1 = No | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD)
Description: Establish MTD of plinabulin in combination with nivolumab and ipilimumab for patients with recurrent SCLC. MTD reflects the highest dose of plinabulin that did not cause a Dose-Limiting Toxicity (DLT) in > 33% of participants. DLTs were defined in accordance to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.
Time Frame: Up to 42 days of first Plinabulin dose
Measure: Number; unit: mg/m^2
Groups:
- Phase I (Dose Escalation): Nivolumab, Ipilimumab and Plinabulin: On Day 1 in a 21-day cycle, all patients will receive nivolumab (1 mg/kg, IV), ipilimumab (3 mg/kg, IV) and plinabulin (escalating cohorts, IV).
  After 4 treatment cycles, ipilimumab will be discontinued and patients will continue treatment with nivolumab 240 mg and plinabulin every 2 weeks (maintenance period) until one of the end of treatment criteria occur.
  Plinabulin escalation is as follows:
  Level -1 : 13.5mg/m^2
  Level 1 (start) : 20mg/m^2
  Level 2 : 30mg/m^2
  Nivolumab: A fully human immunoglobulin (Ig) G4 monoclonal antibody directed against the negative immunoregulatory human cell surface receptor programmed death-1 (PD-1,PCD-1,) with immune checkpoint inhibitory and antineoplastic activities.
  Plinabulin: Plinabulin (BPI-2358) is a synthetic, low molecular weight, new chemical entity originally developed by Nereus Pharmaceuticals, Inc., and now by BeyondSpring Pharmaceuticals, Inc. It belongs to the diketopiperazine class of compounds with a chemical name 2, 5-piperazinedione, 3-[[5-(1,1-dimethylethyl)-1H-imidazol-4-yl[methylene]-6-(phenylmethylene)-, (3Z,6Z) (trivial name t-butyl-dehydrophenylahistin).
  Ipilimumab: Ipilimumab is a monoclonal antibody that works to activate the immune system by targeting CTLA-4, a protein receptor that downregulates the immune system.
Arm/Group | Phase I (Dose Escalation): Nivolumab, Ipilimumab and Plinabulin
Number analyzed (Participants) | 16
mg/m^2 | 30

2. Primary Outcome: Progression-Free Survival (PFS)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease(PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  Progression Free Survival (PFS) is defined as time from registration until disease progression met by RECIST 1.1 or death from any cause.
Time Frame: Up to maximum of 9 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint PFS was defined as all patients with PD-L1 inhibitor resistant recurrent SCLC treated at the plinabulin dose of 30 mg/m^2 with Nivolumab and Ipilimumab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Plinabulin 30mg/m^2 With Nivolumab and Ipilimumab
Number analyzed (Participants) | 27
Months | 1.6 [1.2 to 2.7]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Assess adverse events according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4
Time Frame: Up to a maximum of 43 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for Adverse Events was defined as all patients receiving at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Plinabulin 20mg/m^2 With Nivolumab and Ipilimumab | Plinabulin 30mg/m^2 With Nivolumab and Ipilimumab
Number analyzed (Participants) | 8 | 28
Participants | 8 | 28

4. Secondary Outcome: Number of Participants With Immune-related Adverse Events (irAEs)
Description: Assess Immune-related adverse events according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.
  irAE's are defined as any treatment-related AE that is inflammatory in nature, consistent with the mechanism of action of immunotherapy and generally medically manageable with topical and/or systemic immunosuppressants.
Time Frame: Up to a maximum of 43 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Plinabulin 20mg/m^2 With Nivolumab and Ipilimumab | Plinabulin 30mg/m^2 With Nivolumab and Ipilimumab
Number analyzed (Participants) | 8 | 28
Participants | 1 | 3

5. Secondary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST1.1): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD. Objective Response (OR) = CR + PR
Time Frame: Up to maximum of 9 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Objective Response Rate was defined as all patients with PD-L1 inhibitor resistant recurrent SCLC treated at the plinabulin dose of 30 mg/m^2. Out of 27 PD-L1 inhibitor resistant patients, only 16 were evaluable for ORR.
Measure: Number; unit: Percentage of participants
Arm/Group | Plinabulin 30mg/m^2 With Nivolumab and Ipilimumab
Number analyzed (Participants) | 16
Percentage of participants | 6

6. Secondary Outcome: Clinical Benefit Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD. Clinical Benefit Rate (CBR) = CR+PR+SD per RECIST v1.1.
Time Frame: Up to maximum of 9 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Clinical Benefit Rate was defined as all patients with PD-L1 inhibitor resistant recurrent SCLC treated at the plinabulin dose of 30 mg/m^2. Out of 27 PD-L1 inhibitor resistant patients, only 16 were evaluable for CBR.
Measure: Number; unit: Percentage of participants
Arm/Group | Plinabulin 30mg/m^2 With Nivolumab and Ipilimumab
Number analyzed (Participants) | 16
Percentage of participants | 50

7. Secondary Outcome: Progression Free Survival at 6 Months
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD. PFS is defined as time from registration until disease progression met by RECIST 1.1 or death from any cause. PFS at 6 months is defined as the percentage of patient who was progression free at 6 months from the initiation of treatment.
Time Frame: 6 Months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Progression Free Survival at 6 months was defined as all patients with PD-L1 inhibitor resistant recurrent SCLC treated at the plinabulin dose of 30 mg/m^2 with Nivolumab and Ipilimumab.
Measure: Number; unit: Percentage of participants
Arm/Group | Plinabulin 30mg/m^2 With Nivolumab and Ipilimumab
Number analyzed (Participants) | 27
Percentage of participants | 11

8. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from treatment start until death or date of last contact.
Time Frame: Up to a maximum of 45 months
Population: In accordance with the Statistical Analysis Plan, the analysis population for the endpoint Overall Survival was defined as all patients with PD-L1 inhibitor resistant recurrent SCLC treated at the plinabulin dose of 30 mg/m^2 with Nivolumab and Ipilimumab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Plinabulin 30mg/m^2 With Nivolumab and Ipilimumab
Number analyzed (Participants) | 27
Months | 4.2 [1.9 to 16.9]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 45 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to 43 months.
Arm/Group | Plinabulin 20mg/m^2 With Nivolumab and Ipilimumab | Plinabulin 30mg/m^2 With Nivolumab and Ipilimumab
All-Cause Mortality (participants affected / at risk) | 4/8 | 16/28
Serious Adverse Events (participants affected / at risk) | 4/8 | 21/28
Other Adverse Events (participants affected / at risk) | 8/8 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plinabulin 20mg/m^2 With Nivolumab and Ipilimumab (N=8) | Plinabulin 30mg/m^2 With Nivolumab and Ipilimumab (N=28)
DIARRHEA (GASTROINTESTINAL DISORDERS) | 1 (1) | 0 (0)
FEVER (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 (1) | 0 (0)
HEPATOBILIARY DISORDERS - OTHER, SPECIFY (HEPATOBILIARY DISORDERS) | 1 (1) | 1 (1)
HYPOTENSION (VASCULAR DISORDERS) | 1 (1) | 0 (0)
THROMBOEMBOLIC EVENT (VASCULAR DISORDERS) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (RENAL AND URINARY DISORDERS) | 0 (0) | 1 (1)
ASPIRATION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
BACK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 (0) | 1 (1)
CARDIAC ARREST (CARDIAC DISORDERS) | 0 (0) | 1 (1)
CARDIAC DISORDERS - OTHER, SPECIFY (CARDIAC DISORDERS) | 0 (0) | 1 (1)
COLONIC OBSTRUCTION (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
CONSTIPATION (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
DEATH NOS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (2)
DEHYDRATION (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 1 (2)
DYSPNEA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 3 (4)
EPISTAXIS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
HEMORRHOIDAL HEMORRHAGE (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
HEPATIC FAILURE (HEPATOBILIARY DISORDERS) | 0 (0) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (1)
INVESTIGATIONS - OTHER, SPECIFY (INVESTIGATIONS) | 0 (0) | 1 (1)
KIDNEY INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (1)
LUNG INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 2 (2)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 1 (1)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS)) | 0 (0) | 2 (3)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 2 (3)
PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (1)
PANCREATITIS (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
PLEURAL EFFUSION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 3 (3)
RESPIRATORY FAILURE (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
RESTRICTIVE CARDIOMYOPATHY (CARDIAC DISORDERS) | 0 (0) | 1 (1)
SEIZURE (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
SEPSIS (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (1)
SINUS TACHYCARDIA (CARDIAC DISORDERS) | 0 (0) | 1 (2)
SMALL INTESTINAL OBSTRUCTION (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
SMALL INTESTINAL PERFORATION (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (CARDIAC DISORDERS) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (1)
VASCULAR DISORDERS - OTHER, SPECIFY (VASCULAR DISORDERS) | 0 (0) | 1 (1)
VOMITING (GASTROINTESTINAL DISORDERS) | 0 (0) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plinabulin 20mg/m^2 With Nivolumab and Ipilimumab (N=8) | Plinabulin 30mg/m^2 With Nivolumab and Ipilimumab (N=28)
ABDOMINAL PAIN (GASTROINTESTINAL DISORDERS) | 1 (1) | 2 (3)
ALANINE AMINOTRANSFERASE INCREASED (INVESTIGATIONS) | 2 (3) | 4 (8)
ALKALINE PHOSPHATASE INCREASED (INVESTIGATIONS) | 3 (3) | 6 (8)
ALLERGIC RHINITIS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 0 (0)
ANEMIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 1 (1) | 8 (17)
ANOREXIA (METABOLISM AND NUTRITION DISORDERS) | 2 (2) | 4 (5)
ANXIETY (PSYCHIATRIC DISORDERS) | 1 (1) | 0 (0)
ARTHRALGIA (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 1 (1)
ARTHRITIS (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (INVESTIGATIONS) | 2 (6) | 6 (12)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 3 (20) | 1 (2)
BLOOD BILIRUBIN INCREASED (INVESTIGATIONS) | 1 (1) | 2 (2)
BLURRED VISION (EYE DISORDERS) | 1 (1) | 0 (0)
CARDIAC DISORDERS - OTHER, SPECIFY (CARDIAC DISORDERS) | 1 (1) | 3 (3)
CONSTIPATION (GASTROINTESTINAL DISORDERS) | 1 (1) | 7 (7)
COUGH (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 2 (2) | 3 (3)
DEHYDRATION (METABOLISM AND NUTRITION DISORDERS) | 1 (1) | 3 (3)
DEPRESSION (PSYCHIATRIC DISORDERS) | 1 (1) | 0 (0)
DIARRHEA (GASTROINTESTINAL DISORDERS) | 5 (7) | 9 (11)
DYSPEPSIA (GASTROINTESTINAL DISORDERS) | 1 (1) | 1 (1)
DYSPHAGIA (GASTROINTESTINAL DISORDERS) | 1 (1) | 2 (2)
DYSPNEA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 3 (3) | 5 (6)
ENDOCRINE DISORDERS - OTHER, SPECIFY (ENDOCRINE DISORDERS) | 1 (3) | 0 (0)
FATIGUE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 2 (3) | 10 (13)
FLATULENCE (GASTROINTESTINAL DISORDERS) | 1 (1) | 0 (0)
GAIT DISTURBANCE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 (1) | 1 (1)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (GASTROINTESTINAL DISORDERS) | 1 (1) | 2 (2)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 2 (4) | 5 (7)
GENERALIZED MUSCLE WEAKNESS (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 1 (1)
HEADACHE (NERVOUS SYSTEM DISORDERS) | 3 (4) | 3 (5)
HEMOGLOBIN INCREASED (INVESTIGATIONS) | 1 (2) | 0 (0)
HYPERGLYCEMIA (METABOLISM AND NUTRITION DISORDERS) | 2 (4) | 4 (4)
HYPERTENSION (VASCULAR DISORDERS) | 1 (1) | 7 (11)
HYPERTHYROIDISM (ENDOCRINE DISORDERS) | 2 (2) | 0 (0)
HYPOGLYCEMIA (METABOLISM AND NUTRITION DISORDERS) | 1 (4) | 2 (3)
HYPOKALEMIA (METABOLISM AND NUTRITION DISORDERS) | 3 (4) | 5 (6)
HYPOMAGNESEMIA (METABOLISM AND NUTRITION DISORDERS) | 1 (1) | 4 (5)
HYPONATREMIA (METABOLISM AND NUTRITION DISORDERS) | 3 (3) | 4 (4)
HYPOPHOSPHATEMIA (METABOLISM AND NUTRITION DISORDERS) | 1 (1) | 1 (1)
HYPOTHYROIDISM (ENDOCRINE DISORDERS) | 1 (1) | 2 (2)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (INFECTIONS AND INFESTATIONS) | 1 (1) | 1 (1)
INFUSION RELATED REACTION (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 3 (3) | 8 (17)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 1 (1) | 0 (0)
INSOMNIA (PSYCHIATRIC DISORDERS) | 2 (2) | 2 (3)
LIPASE INCREASED (INVESTIGATIONS) | 1 (3) | 4 (4)
LUNG INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1) | 3 (3)
LYMPHOCYTE COUNT DECREASED (INVESTIGATIONS) | 3 (3) | 8 (14)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (2) | 2 (2)
NAUSEA (GASTROINTESTINAL DISORDERS) | 5 (11) | 15 (25)
NECK EDEMA (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 (2) | 0 (0)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (NERVOUS SYSTEM DISORDERS) | 1 (1) | 1 (1)
NON-CARDIAC CHEST PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 (1) | 3 (5)
ORAL PAIN (GASTROINTESTINAL DISORDERS) | 1 (1) | 0 (0)
PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 4 (4) | 5 (5)
PAIN IN EXTREMITY (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1) | 1 (1)
PLATELET COUNT DECREASED (INVESTIGATIONS) | 2 (2) | 4 (8)
POSTNASAL DRIP (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 0 (0)
PRURITUS (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (6) | 5 (5)
PSYCHIATRIC DISORDERS - OTHER, SPECIFY (PSYCHIATRIC DISORDERS) | 1 (1) | 0 (0)
RASH MACULO-PAPULAR (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 2 (2) | 4 (4)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 2 (2)
SEIZURE (NERVOUS SYSTEM DISORDERS) | 1 (1) | 0 (0)
SERUM AMYLASE INCREASED (INVESTIGATIONS) | 1 (1) | 2 (2)
SINUS TACHYCARDIA (CARDIAC DISORDERS) | 1 (1) | 1 (1)
SORE THROAT (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1) | 0 (0)
UPPER RESPIRATORY INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1) | 0 (0)
VOMITING (GASTROINTESTINAL DISORDERS) | 3 (6) | 14 (25)
WEIGHT GAIN (INVESTIGATIONS) | 1 (1) | 0 (0)
WHITE BLOOD CELL DECREASED (INVESTIGATIONS) | 2 (4) | 6 (10)
ACIDOSIS (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 1 (1)
ALOPECIA (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 1 (1)
ASPIRATION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
BACK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 (0) | 4 (4)
CARDIAC TROPONIN I INCREASED (INVESTIGATIONS) | 0 (0) | 1 (1)
CARDIAC TROPONIN T INCREASED (INVESTIGATIONS) | 0 (0) | 3 (3)
CHEST PAIN - CARDIAC (CARDIAC DISORDERS) | 0 (0) | 1 (1)
CHILLS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (1)
COLITIS (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
CONFUSION (PSYCHIATRIC DISORDERS) | 0 (0) | 1 (1)
CREATININE INCREASED (INVESTIGATIONS) | 0 (0) | 2 (3)
DEATH NOS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (1)
DENTAL CARIES (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
DRY SKIN (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 1 (1)
DYSARTHRIA (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
DYSGEUSIA (NERVOUS SYSTEM DISORDERS) | 0 (0) | 3 (3)
EDEMA FACE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 0 (0) | 1 (1)
FEVER (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 0 (0) | 3 (5)
FLUSHING (VASCULAR DISORDERS) | 0 (0) | 2 (2)
GASTROPARESIS (GASTROINTESTINAL DISORDERS) | 0 (0) | 1 (1)
HICCUPS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
HOARSENESS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
HYPERCALCEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 2 (2)
HYPERMAGNESEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 1 (1)
HYPERNATREMIA (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 1 (2)
HYPOALBUMINEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 2 (3)
HYPOCALCEMIA (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 3 (3)
HYPOTENSION (VASCULAR DISORDERS) | 0 (0) | 3 (5)
HYPOXIA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
IMMUNE SYSTEM DISORDERS - OTHER, SPECIFY (IMMUNE SYSTEM DISORDERS) | 0 (0) | 2 (2)
LETHARGY (NERVOUS SYSTEM DISORDERS) | 0 (0) | 2 (2)
LEUKOCYTOSIS (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 0 (0) | 1 (1)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (METABOLISM AND NUTRITION DISORDERS) | 0 (0) | 2 (3)
MUCOSITIS ORAL (GASTROINTESTINAL DISORDERS) | 0 (0) | 2 (2)
MUSCLE WEAKNESS LEFT-SIDED (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 (0) | 1 (1)
MUSCLE WEAKNESS UPPER LIMB (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (CARDIAC DISORDERS) | 0 (0) | 1 (1)
NEUTROPHIL COUNT DECREASED (INVESTIGATIONS) | 0 (0) | 2 (3)
PARESTHESIA (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (2)
PLEURAL EFFUSION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 2 (4)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (RENAL AND URINARY DISORDERS) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 0 (0) | 1 (1)
SEPSIS (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (1)
SINUS BRADYCARDIA (CARDIAC DISORDERS) | 0 (0) | 1 (1)
SINUS PAIN (NERVOUS SYSTEM DISORDERS) | 0 (0) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 4 (5)
SKIN ULCERATION (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 0 (0) | 1 (1)
SYNCOPE (NERVOUS SYSTEM DISORDERS) | 0 (0) | 3 (4)
THROMBOEMBOLIC EVENT (VASCULAR DISORDERS) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (INFECTIONS AND INFESTATIONS) | 0 (0) | 1 (1)
WEIGHT LOSS (INVESTIGATIONS) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/93/NCT03575793/Prot_SAP_000.pdf